CLINICAL TRIAL: NCT05624034
Title: To Study the Electrogastrography [EGG]Abnormalities in Healthy Subjects and in Patients With Idiopathic and Diabetic Gastroparesis: A Prospective Single Center Study.
Brief Title: To Study the EGG Abnormalities in Healthy Subjects and in Patients With Idiopathic and Diabetic Gastroparesis.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Rakesh Kalapala, Director Endoscopy[ Center for obesity and metabolic therapy], Asian Institute of Gastroenterology, India
Other Study IDs: AIG/IEC-BH&R32/07.2022-03
Record Dates: First submitted 2022-11-14; First posted 2022-11-21 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Gastroparesis; Diabetes Complications; Idiopathic Gastric Motility Disorder; Dyspepsia
Keywords: gastroparesis; dyspepsia; gastric myoelectric activity
MeSH Terms: conditions — Gastroparesis; Diabetes Complications; Dyspepsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- Healthy group: Subjects with no previous medical history (healthy volunteers) will be assessed for eligibility criteria.
  Interventions: Device: Electrogastrography
- Idiopathic Gastroparesis: Patients with symptoms of Gastroparesis based on ROME IV criteria and not having a known cause of gastroparesis like endocrine, neurological, rheumatological disorder.
  Interventions: Device: Electrogastrography
- Diabetic Gastroparesis: Patients with symptoms of Gastroparesis based on ROME IV criteria and Diabetes mellitus of any duration.
  Interventions: Device: Electrogastrography

INTERVENTIONS:
Device: Electrogastrography — Electrogastrography is used to study abnormalities in healthy subjects and in patients with Diabetic and Idiopathic Gastroparesis

SUMMARY:
Electrogastrogram (EGG) is a non-invasive method for recording myoelectric activities by placing electrodes on the abdomen surface. Many studies suggested EGG measures the gastric slow wave frequency effectively; the relative change in EGG signal amplitude would reflect the contractility of the stomach. Thus, this technique is used to study the pathophysiological processes of diseases such as functional dyspepsia and many more .

The present study aims to study the EGG pattern in healthy individuals in Indian population and the factors associated with it.

DETAILED DESCRIPTION:
Electrogastrogram [EGG] is an authentic method to detect gastrointestinal diseases accompanied by gastric motility abnormalities . The present study would help to determine the normatic values of EGG in healthy population and EGG changes in patients with idiopathic gastroparesis. This pilot study would provide findings/abnormalities seen in study population and may be helpful in providing a comparative data for proper treatment and a better quality of life patients suffering from dyspepsia.

All the eligible subjects will undergo study procedure i.e. EGG. The study procedure will conduct as per standard study protocol. EGG is a non-invasive, painless method for the measurement of gastric myoelectrical activity. EGG takes around two hours to complete the procedure and no side effects reported. Following steps are included in the procedure

* Subject lie on back on a procedure table.
* Investigator or technician tapes electrodes to Subject's abdomen (belly). The electrodes are similar to those used for other tests, such as an ECG (electrocardiogram). The electrodes measure electrical signals coming from stomach muscles. They send the signals to a computer that records the signals as a graph.
* Investigator or technician records a test while Subject's stomach is empty. An hour later, Subject have something to eat and drink. Investigator or technician then records a second test. The test and electrodes are painless.
* The electrodes are removed. EGG test is completed at this point.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet the following criteria to be included in the study:
* Healthy subjects 20 Males and 20 females subjects atleast one will be taken from each group [18-20,20-30,30-40,40-50,50-60,60-70yrsAbsence of previous upper gastrointestinal surgery anytime in past.
* Absence of drugs which affect the upper gastrointestinal system in 3 months.
* Absence of diabetes,thyroid disorder or neuromuscular disorder.
* Subject who has read the informed consent form, has understood the relevant aspects of the study, and grants his/her authorization to participate by signing the informed consent form before the inclusion in the study and the performance of any procedure
* Subject willing to use appropriate method of contraception as per investigator's discretion, throughout the study
* Idiopathic Gastroparesis
* Male and female subjects above 18 to 70 years of age.
* Subject who has read the informed consent form, has understood the relevant aspects of the study, and grants his/her authorization to participate by signing the informed consent form before the inclusion in the study and the performance of any procedure
* Subject willing to use appropriate method of contraception as per investigator's discretion, throughout the study
* Patient's having symptoms of dyspepsia based on ROME IV Criteria and not having a known cause of gastroparesis like endocrine, neurological, rheumatological disorder.
* ROME IV criteria for Functional Dyspepsia* (Diagnostic criteria**): One or more of the following
* Bothersome postprandial fullness
* Bothersome early satiation
* Bothersome epigastric pain
* Bothersome epigastric burning AND
* No evidence of structural disease (including at upper endoscopy) that is likely to explain the symptoms

  -*Must fulfill criteria for Postprandial Distress Syndrome (PDS) and/or Epigastric Pain Syndrome (EPS)

  -**Criteria fulfilled for the last 3 months with symptom onset at least 6 months prior to diagnosis
* Diabetic Gastroparesis
* Male and female subjects above 18 to 70 years of age.
* Subject who has read the informed consent form, has understood the relevant aspects of the study, and grants his/her authorization to participate by signing the informed consent form before the inclusion in the study and the performance of any procedure
* Subject willing to use appropriate method of contraception as per investigator's discretion, throughout the study
* Patient's having symptoms of dyspepsia based on ROME IV Criteria and Diabetes mellitus of any duration

Exclusion Criteria:

* Subjects who meet any of the following criteria will be excluded from the study:
* For Idiopathic Gastroparesis
* Subjects suffering from Diabetes
* Subjects with history of any bariatric procedures/ gastric surgeries in the past
* Females who are pregnant
* Subjects taking following medications within 72 hours to the start of the study: Opioids, TCA, Calcium channel blockers, anti-psychotics, anti-cholinergic, steroids, L-Dopa
* Subjects with electrolyte abnormalities like hypokalaemia, hypomagnesemia
* Subjects with known cases of thyroid disorder (hypo or hyperthyroidism)
* Subjects who are unsuitable for any other reason to participate in the study in the opinion of the investigator
* For Diabetic Gastroparesis
* Subjects with history of any bariatric procedures/ gastric surgeries in the past
* Females who are pregnant
* Subjects taking following medications within 72 hours to the start of the study: Opioids, TCA, Calcium channel blockers, anti-psychotics, anti-cholinergic, steroids, L-Dopa
* Subjects with electrolyte abnormalities like hypokalaemia, hypomagnesemia
* Subjects with known cases of thyroid disorder (hypo or hyperthyroidism)
* Subjects who are unsuitable for any other reason to participate in the study in the opinion of the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 40 healthy individuals, 50 diabetic gastroparesis patients and 50 idiopathic gastroparesis will be enrolled in the study as per the inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
EGG findings | 6 months
  To study the EGG abnormalities in healthy subjects and in patients with Diabetic and Idiopathic Gastroparesis

SECONDARY OUTCOMES:
Factors affecting the condition | 6 months
  To study factors associated with abnormalities noted in EGG

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh Kalapala, MBBS,MD,DM, Study Director — Senior consultant
Locations (1):
- AIG Hospitals, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Riezzo G, Russo F, Indrio F. Electrogastrography in adults and children: the strength, pitfalls, and clinical significance of the cutaneous recording of the gastric electrical activity. Biomed Res Int. 2013;2013:282757. doi: 10.1155/2013/282757. Epub 2013 May 25. PMID 23762836
- [Background] Al Kafee A, Akan A. Analysis of gastric myoelectrical activity from the electrogastrogram signals based on wavelet transform and line length feature. Proc Inst Mech Eng H. 2018 Apr;232(4):403-411. doi: 10.1177/0954411918757812. Epub 2018 Feb 14. PMID 29441814

DOCUMENTS (1):
  • Study Protocol (2022-07-29): https://cdn.clinicaltrials.gov/large-docs/34/NCT05624034/Prot_000.pdf